CLINICAL TRIAL: NCT01325025
Title: Study of the Natural History of Cerebral White Matter Involvement in Metachromatic Leukodystrophy, Using High-field MRI and Diffusion Tensor Imaging
Brief Title: Imaging Study of the White Matter Lesions in Children With Metachromatic Leucodystrophy
Acronym: HCIT-MLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Leukodystrophy Association (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P071232
Record Dates: First submitted 2011-03-09; First posted 2011-03-29 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Late Infantile Metachromatic Leukodystrophy
Keywords: Metachromatic Leukodystrophy; Demyelinating Diseases; Magnetic Resonance Imaging; Diffusion Tensor Imaging; Relaxometry; Spectroscopy; Longitudinal Studies
MeSH Terms: conditions — Leukodystrophy, Metachromatic; Demyelinating Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Other): Patients with a metachromatic leukodystrophy
  Interventions: Other: High-field MRI (3 Teslas)
- Control (Other): Epileptic population
  Interventions: Other: High-field MRI (3 Teslas)

INTERVENTIONS:
Other: High-field MRI (3 Teslas) — * anatomical location
  * conventional anatomical sequence T1, T2, FLAIR
  * diffusion tensor sequence (21 directions)
  * high angular resolution diffusion (HARDI) sequence
  * field map
  * reflexology T1, T2
  * spectroscopic imaging sequence
  Arms: Patients
Other: High-field MRI (3 Teslas) — * anatomical location
  * conventional anatomical sequence T1, T2, FLAIR
  * diffusion tensor sequence (21 directions)
  * high angular resolution diffusion (HARDI) sequence
  * field map
  * reflexology T1, T2
  * spectroscopic imaging sequence
  Arms: Control

SUMMARY:
High-field MRI and diffusion tensor imaging with 3D reconstruction of the myelin tracks, in combination with multivoxel proton spectroscopy, will allow to precise more accurately the evolution of the white matter lesions in patients affected with Metachromatic Leukodystrophy (particularly in the initial phase of the disease). This will increase the knowledge of the disease and provide new indicators for the selection and evaluation of patients eligible for new therapeutic approaches.

DETAILED DESCRIPTION:
Metachromatic Leukodystrophy (MLD) is a rare autosomal recessive disorder caused by the deficiency of the Arylsulfatase A enzyme (ARSA), resulting in accumulation of galactosyl sulfatide (cerebroside sulfate), a major constituent of the myelin sheath. Accumulation of sulfatides leads to a progressive degeneration of the white matter in the central and peripheral nervous systems (CNS, PNS) and to a neuronal degeneration. The late-infantile form of MLD, which is usually diagnosed in the second year of life, is the most frequent and severe form of the disease. The prognosis is severe, leading to vegetative stage or death within few years after the diagnosis. There is no treatment for patients affected with this early-onset form of the disease.

Conventional MRI (1.5 Tesla) shows extensive involvement of the cerebral white matter (hypo-T1, hyper- T2 and FLAIR signals) indicative of rapidly progressing leukodystrophy. Early cortical atrophy reflects associated neuronal involvement. Proton MR spectroscopy demonstrates abnormalities of choline and N-acetyl-aspartate (demyelination, neuronal loss), which are non-specific but can serve as indicators to monitor the effects of any therapeutic intervention.

In early-onset forms of MLD, conventional MRI becomes abnormal at a relatively advanced stage of the disease and the neuroradiological diagnosis may be difficult before the age of 2 - 2 1/2 years of age. Moreover, topography and extent of detectable lesions are poorly correlated with the disease severity.

In order to improve information provided by neuroimaging, this study aims to investigate prospectively and longitudinally (over a period of 6 months) white and grey matter lesions in 10 MLD children aged 1 to 6 years, using high-field MRI (3 Teslas) and diffusion tensor imaging (DTI) with 3D reconstruction of the myelin tracks. The time interval between diagnosis and inclusion will not exceed 18 months, thus patients will be included at an early stage of their disease. Each time-point (T0 and 6 months) will also include neurological evaluation to correlate the imaging, cognitive and motor functions. Children will be included over a period of 5 years. The total duration of the study will be 5.5 years. Controls will include 25 age-matched children with cryptogenic partial epilepsy who should have a high-field MRI to detect structural abnormalities. Controls will have a MRI and cognitive evaluation at T0 and 12 months if necessary. This study will increase our knowledge of the natural history of MLD and provide new indicators for the selection and evaluation of patients eligible for new therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria (patients):

* Children with proven metachromatic leukodystrophy (MLD) with decreased activity of arylsulfatase A enzyme in leukocytes and abnormal excretion of urinary sulfatides
* Age ≥ 1 year and ≤ 6 years
* Recently diagnosed (within < 18 months)

Inclusion Criteria (control):

* Children with partial cryptogenic epilepsy or with a suspected brain lesion on conventional MRI, who should have high-field MRI to detect structural abnormalities that could benefit from surgical resection
* Age ≥ 1 year and ≤ 6 years

Exclusion Criteria:

* Evolutive heart, pulmonary, renal or gastrointestinal disease
* Contra-indication to sedation
* Contra-indication to MRI (implanted magnetic material)

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2010-11; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assess the natural history of the white matter and cortex lesions in MLD using diffusion tensor imaging (DTI)and relaxometry/ high field MRI. | At inclusion (T0) and 12 months for control. At T0 then at 6 months for patients
  The following parameters will be studied: quantitative measurements of mean diffusivity, longitudinal and transverse fractional anisotropy in ROIs (regions of interest), 3D-tractographic reconstruction of the myelin tracks.

SECONDARY OUTCOMES:
Assess the natural history of the white matter and cortex lesions in MLD using using multi-voxel spectroscopic imaging. | At inclusion (T0) and 12 months for control. At T0 then at 6 months for patients
Assess the evolution of cortical atrophy, | At inclusion (T0) and 12 months for control. At T0 then at 6 months for patients
Correlate the neuroimaging parameters with motor function measure (Gross Motor Function Measure) and cognitive tests (BSID, WPPSI). | At inclusion (T0) and 12 months for control. At T0 then at 6 months for patients

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Sevin, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (3):
- France (3):
  - Unité de recherche biomédicale, Neurospin, I2BM / DSV / SAC/ CEA,, Gif-sur-Yvette
  - Service de Neurologie Pédiatrique, Hôpital Bicêtre, Paris
  - Bâtiment Lavoisier - Unité INSERM U 663,Hôpital Necker Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No